CLINICAL TRIAL: NCT01954355
Title: LDE225 in Combination With Paclitaxel in Patients With Advanced Solid Tumors - A Multicenter Phase I Trial
Brief Title: LDE225 and Paclitaxel in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 65/12; CLDE225XCH01T (Other: Novartis); 2013DR1122 (Other: Swissmedic); SNCTP000001101 (Other: SNCTP)
Record Dates: First submitted 2013-09-19; First posted 2013-10-01 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Solid Tumor; Ovarian Cancer
Keywords: advanced solid tumor; ovarian cancer; LDE225; Paclitaxel; Hedgehog inhibitor
MeSH Terms: conditions — Ovarian Neoplasms | interventions — sonidegib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LDE225 & Paclitaxel (Experimental): Phase I, Part A: LDE225: dose escalation in cohorts of 3-6 patients (days 1-28) and Paclitaxel 80 mg/m2 (days 1, 8, 15)
  Phase I, Part B and C: LDE225: RP2D established in Part A (days 1-28) and Paclitaxel 80 mg/m2 (days 1, 8, 15)
  Interventions: Drug: LDE225; Drug: Paclitaxel

INTERVENTIONS:
Drug: LDE225 — 400, 600 and 800 mg OD
Drug: Paclitaxel — 80 mg/m2 (days 1, 8, 15)
  Other Names: Taxol

SUMMARY:
The primary aim of this trial is to establish the maximum tolerated dose (MTD) and the recommended phase II dose (RP2D) of LDE225 given in combination with standard doses of paclitaxel in patients with advanced solid tumors. In addition, the preliminary anti-tumor activity of this combination will be assessed, in particular in ovarian cancer.

DETAILED DESCRIPTION:
This is a multicenter, open label phase I dose-escalation trial of LDE225 administered once daily (OD) with Paclitaxel administered weekly for three weeks (days 1, 8, 15) in 28-day cycles in adult patients with advanced solid tumors that have progressed despite standard therapy.

The trial will consist of three parts. In Part A (dose escalation following a standard 3+3 design), patients with previously treated advanced solid tumors will receive escalating doses of LDE225 in combination with standard Paclitaxel doses, to define the MTD and the RP2D of LED225 OD that can be given in combination with standard doses of Paclitaxel. Once the MTD and RP2D is established in 6 patients, then part B will start.

Part B and C are expansion cohorts in patients with advanced platinum-resistant ovarian cancer (6 patients each) to further evaluate the safety of the combination and to assess for any preliminary antitumor activity.

In Part B, any prior taxane therapy must have been administered on a 3-week schedule. In Part C, prior taxane therapy must have been administered on weekly schedule and has to be followed by a wash-out period of at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must give written informed consent before registration.
* For Part A: Histologically or cytologically confirmed diagnosis of advanced solid tumors that have progressed despite standard therapy. No more than two prior lines of chemotherapy for advanced disease.
* For Part B: Histologically or cytologically confirmed diagnosis of advanced ovarian cancer. Prior chemotherapy must have contained a platinum and a taxane at some point. Any prior taxane therapy must have been administered on a 3-week schedule. A maximum of 2 prior chemotherapy lines for advanced disease will be permitted. Patients must be refractory (PD during chemotherapy) or resistant (PD within 6 months of completing chemotherapy) to their last platinum-containing chemotherapy regimen.
* For Part C: Histologically or cytologically confirmed diagnosis of advanced ovarian cancer. Prior chemotherapy must have contained a platinum and a taxane at some point. Prior taxane therapy must have been administered on weekly schedule and must be followed by a wash-out period of at least 6 months. A maximum of 2 prior chemotherapy lines for advanced disease will be permitted. Patients must be refractory (PD during chemotherapy) or resistant (PD within 6 months of completing chemotherapy) to their last platinum-containing chemotherapy regimen.
* For Parts B and C, patients must have measurable disease according to RECIST v1.1 Radiological evaluations to be performed within 4 weeks before registration.
* WHO performance status 0-1
* Age ≥ 18 years
* Hematological values: ANC ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, Hemoglobin ≥ 100 g/L
* Adequate hepatic function: bilirubin ≤ 1.5 x ULN, AST and ALT ≤ 2.5 x ULN or ≤ 5.0 x ULN if liver metastases are present
* Creatine phosphokinase (CPK) ≤ ULN
* Albumin ≥ 30g/L
* Adequate renal function (calculated creatinine clearance > 50 mL/min, according to the formula of Cockcroft-Gault, see Appendix 3)
* Archived tumor tissue must be available.
* Women are not breastfeeding.
* Women of child-bearing potential are using effective contraception, are not pregnant and agree not to become pregnant during participation in the trial and during the 12 months thereafter. They are required to have a negative serum pregnancy test before registration (within 7 days).
* Men agree not to father a child during participation in the trial and during 12 months thereafter. They agree to use effective contraception.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the trial or those who prior to the first dose of combination have not recovered to ≤ CTCAE Grade 1 from adverse events due to agents administered more than 4 weeks earlier
* Symptomatic brain metastases
* Prior therapy with a Hedgehog inhibitor
* Known or prior hypersensitivity to taxanes or drugs containing Cremophor in spite of premedication
* Positive HIV test
* Positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test
* Impairment of gastrointestinal (GI) function or GI disease (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Impaired cardiac function or clinically significant heart disease
* Patients who are receiving treatment with medications that are known to be strong inhibitors or inducers of CYP3A4/5 or drugs metabolized by CYP2B6 or CYP2C9 that cannot be discontinued
* Patients who are currently receiving treatment with warfarin sodium (Coumadin)
* Patients who are currently receiving immunosuppressive treatment and in whom the treatment cannot be discontinued prior to starting trial drug.
* Patients receiving medications that are recognized to cause rhabdomyolysis, such as HMG CoA reductase inhibitors (statins) clofibrate, gemfibrozil, and that cannot be stopped at least 2 weeks prior to the initiation of LDE225 treatment
* Patients who have undergone major surgery ≤ 2 weeks prior to starting trial drug or who have not recovered from such therapy
* Psychiatric disorder precluding understanding of information on trial related topics, giving informed consent, or interfering with compliance for oral drug intake.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) of the combination of LDE225 with paclitaxel in patients with advanced solid tumors | until up to 4 weeks after start of trial therapy

SECONDARY OUTCOMES:
Frequency and severity of adverse events based on the Common Terminology Criteria for Adverse Events V.4.0 (CTCAE). | expected average 3 months
Objective tumor responses based on RECIST 1.1 criteria. | expected average 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios Stathis, MD, Study Chair — IOSI, Ospedale San Giovanni; Cristiana Sessa, Prof Dr med, Study Chair — IOSI, Ospedale San Giovanni
Locations (4):
- Switzerland (4):
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Kantonsspital Graubünden, Chur
  - Centre Pluridisciplinaire d'Oncologie CHUV, Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No